CLINICAL TRIAL: NCT05465369
Title: Clinical Assessment of Injectable Flowable Composite with Giomer Based Technology Versus High Viscosity Glass Ionomer Restorations in Atraumatic Restorative Treatment (ART) for Cancer Patients (One Year Randomized Clinical Trial)
Brief Title: Clinical Assessment of Injectable Flowable Composite with Giomer Technology Vs High Viscosity Glass Ionomer Restorations in ART for Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Principal Investigator, Mennatallah Ahmed Shawkey, Master's degree student ,faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPR 14/8/2022
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-02

CONDITIONS: Secondary Caries; Fracture Tooth; Discoloration, Tooth
Keywords: Tooth Caries; Discoloration, Tooth
MeSH Terms: conditions — Tooth Fractures; Tooth Discoloration; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- injectable flowable composite with giomer technology (beatifil flow plus x) (Experimental): Injectable flowable Giomer composites is a material used for direct filling techniques has been developed over the past years. It has the property of Giomer technology that able to release and recharge fluoride and other beneficial ions for the life of the restoration and induce remineralization of the underlying hard dental tissues . Injectable flowable Giomer composite (Beautifil flow plus x) has a long-term clinical performance like conventional composite., it also aids in decrease acid production and formation of antiacid resistant layer, help in reduction of tooth mineral solubility also it has high survival rate and wear resistance in high stress bearing areas in posterior teeth Beautifil Flow Plus X also helps to remineralise the tooth structure for sustainable caries prevention and easily polishes for long-lasting luster
  Interventions: Other: giomer
- high viscosity glass ionomer (Equia Fil ) in ART (Active Comparator): High viscous glass ionomer, the most suitable restorative material for ART procedure and can be used outside the dental clinic, which increases the opportunity for dental care , using a high-viscosity glass-ionomer as an ART sealant in both primary and permanent posterior teeth have a high caries preventive effect High viscosity glass ionomer (EQUIA Fil) has new technology involves ultrafine, and highly reactive glass diffused within the glass-ionomer fillers to increase and enhance matrix formation. This system allows ion availability and builds a stronger matrix structure with greater physical properties, wear resistance and fluoride release. Mechanical properties and fluoride release is the most important features to evaluate glass ionomer restorative material and it's proven that EQUIA Fil fulfilled all these requirement
  Interventions: Other: high viscosity glass ionomer

INTERVENTIONS:
Other: giomer — injectable flowable Giomer composites is a material used for direct filling techniques has been developed over the past years. It has the property of Giomer technology that able to release and recharge fluoride and other beneficial ions for the life of the restoration and induce remineralization of the underlying hard dental tissues . Injectable flowable Giomer composite (Beautifil flow plus x) has a long-term clinical performance like conventional composite., it also aids in decrease acid production and formation of antiacid resistant layer, help in reduction of tooth mineral solubility also it has high survival rate and wear resistance in high stress bearing areas in posterior teeth Beautifil Flow Plus X also helps to remineralise the tooth structure for sustainable caries prevention and easily polishes for long-lasting luster
  Other Names: Beautifil Flow Plus X
  Arms: injectable flowable composite with giomer technology (beatifil flow plus x)
Other: high viscosity glass ionomer — High viscous glass ionomer, the most suitable restorative material for ART procedure and can be used outside the dental clinic, which increases the opportunity for dental care , using a high-viscosity glass-ionomer as an ART sealant in both primary and permanent posterior teeth have a high caries preventive effect High viscosity glass ionomer (EQUIA Fil) has new technology involves ultrafine, and highly reactive glass diffused within the glass-ionomer fillers to increase and enhance matrix formation. This system allows ion availability and builds a stronger matrix structure with greater physical properties, wear resistance and fluoride release. Mechanical properties and fluoride release is the most important features to evaluate glass ionomer restorative material and it's proven that EQUIA Fil fulfilled all these requirement
  Other Names: Equia fill
  Arms: high viscosity glass ionomer (Equia Fil ) in ART

SUMMARY:
Aim of the Study:

This study will compare between injectable flowable composite (Beautifil flow plus x) and high viscosity glass ionomer (Equia Fil) by ART caries preventive protocol in high caries risk patients receiving chemotherapy and/or radiotherapy

DETAILED DESCRIPTION:
Statement of the problem:

Chemotherapy and radiation therapy may cause changes in the lining of the mouth and the salivary glands. This can upset the healthy balance of bacteria. These changes may lead to mouth sores, infections, and tooth decay.

Rationale:

Patients under chemotherapy treatment and radiotherapy are systemically compromised and undergo hospital manipulations and residency, increasing their caries risk, fear, and anxiety. That's why they need specific caries preventive protocols designed for high-risk patients. Atraumatic restorative treatment (ART) is recommended for these patients to decrease pain and anxiety.

Atraumatic restorative treatment (ART) and interim therapeutic restoration (ITR) have had increased interest in the past few years. ART and ITR are comparative approaches and are performed utilizing the same material, but they contrast within the reason of their utilize. ART is very effective as a restorative technique since it is more conservative than conventional treatment. Also in this technique, we avoid using rotary equipment and dental anaesthesia, which increase anxiety during the dental procedure. ITR, on the other hand, is used as a temporary restoration that will be replaced with a more definitive one.

Injectable flowable Giomer composites are a material used for direct filling techniques has been developed over the past years. It has the property of Giomer technology that is able to release and recharge fluoride and other beneficial ions for the life of the restoration and induce remineralization of the underlying hard dental tissues. Injectable flowable Giomer composite (Beautiful flow plus x) has a long-term clinical performance like conventional composite., it also aids in decreasing acid production and formation of an antiacid resistant layer, helps in the reduction of tooth mineral solubility also has a high survival rate and wear resistance in high stress-bearing areas in posterior teeth.

Beautiful Flow Plus X also helps to remineralise the tooth structure for sustainable caries prevention and easily polishes for long-lasting lustre

ELIGIBILITY:
Inclusion Criteria:

* existing caries in permanent posterior teeth
* Permanent posterior teeth with active carious lesion class I and class II without any signs and symptoms of pulp disease.
* Teeth in normal occlusion
* Absence of any active periodontal disease.

Exclusion Criteria:

* Patients whose systemic involvement was too advanced to allow dental manipulation, such as those who were admitted to the intensive care unit
* Patients with parafunctional habits
* Presence of any sign or symptoms of irreversible Pulpitis or necrotic pulp
* Partially erupted teeth

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
recurrence of caries | 12 months
  Modified USPHS criteria

SECONDARY OUTCOMES:
Restoration clinical performance | 12 months
  Color match Alfa: no change in color Bravo: change in color Marginal discoloration Alfa: no discoloration bravo: discoloration for less than one - half of the margins Charlie: discoloration for more than one -half of margin Relapse of caries Alfa: no caries present Charlie: caries present Anatomical shape Alfa: clinically ideal Bravo: clinically acceptable Charlie: clinically unacceptable Marginal integrity Alfa: Closely adapted, no visible crevice Bravo: Visible crevice, explorer will penetrate Surface texture Alfa: no defect Bravo: minimal defects Charlie: severe defects rest of modified usphs criteria

CONTACTS AND LOCATIONS:
Overall Officials: menna ahmed shawkey, masters, Principal Investigator — Cairo University; Rawda Hisham abd elaziiz, Study Chair — Cairo University
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, El Sayeda Zeinab, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Aim of the Study:
  This study will compare between injectable flowable composite (Beautifil flow plus x) and high viscosity glass ionomer (Equia Fil) by ART caries preventive protocol in high caries risk patients receiving chemotherapy and/or radiotherapy.
Supporting Information: Study Protocol
Time Frame: the restoration will be evaluated at T0: Baseline T1: 6 months measurement. T2: 12 months measurement.
Access Criteria: Young adult (12-18) years Patients who have existing caries in permanent posterior teeth Teeth inclusion criteria Permanent posterior teeth with active carious lesion class I and class II without any signs and symptoms of pulp disease.
  Teeth in normal occlusion Absence of any active periodontal disease.